CLINICAL TRIAL: NCT04551118
Title: Efficacy of Transcranial Electrical Stimulation (tES) of Dorsolateral- Prefrontal Cortex on Emotion Processing: A Randomized, Single-blind, Sham-controlled Trial
Brief Title: Efficacy of Transcranial Electrical Stimulation (tES) on Emotion Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: tES-2019-TJAH
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: transcranial Electrical Stimulation (tES)
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tACS group (Experimental): Participants receive 20 min sessions of 1.5 mA alternating current delivered over the dorsolateral prefrontal cortex, for 7 consecutive days.
  Interventions: Device: Transcranial alternating current stimulation (tACS) -active
- tDCS group (Experimental): Participants receive 20 min sessions of 1.5 mA direct current delivered over the dorsolateral prefrontal cortex, for 7 consecutive days.
  Interventions: Device: Transcranial direct current stimulation (tDCS)-active
- Sham group (Sham Comparator): Participants receive sham stimulation that administered similarly, but with current continued less than 30s.
  Interventions: Device: Transcranial electrical stimulation (TES)-sham

INTERVENTIONS:
Device: Transcranial alternating current stimulation (tACS) -active — Transcranial alternating current stimulation (tACS) is a non-invasive neuromodulation technique of the brain with an AC micro-electrical stimulator, two rubber electrodes in saline-soaked sponges, and a control software to set the output of the stimulation type. Participants receive 20 min sessions of 1.5 mA alternating current delivered over the dorsolateral prefrontal cortex, for 7 consecutive days.
  Other Names: tACS active
  Arms: tACS group
Device: Transcranial direct current stimulation (tDCS)-active — Transcranial direct current stimulation (tDCS) is a non- invasive neuromodulation technique of the brain with a DC micro-electrical stimulator, two rubber electrodes in saline-soaked sponges, and a control software to set the output of the stimulation type. Participants receive 20 min sessions of 1.5 mA direct current delivered over the dorsolateral prefrontal cortex, for 7 consecutive days.
  Other Names: tDCS active
  Arms: tDCS group
Device: Transcranial electrical stimulation (TES)-sham — Transcranial electrical stimulation (TES) is a non-invasive neuromodulation technique of the brain with micro-electrical stimulator, two rubber electrodes in saline-soaked sponges, and a control software to set the output of the stimulation type. Participants receive sham stimulation over the dorsolateral prefrontal cortex, with current turned off after 30 second. The session last 20 min for 7 consecutive days.
  Arms: Sham group

SUMMARY:
The aim of this study is to assess the efficacy of transcranial Electrical Stimulation (tES) on emotion processing of healthy participants. Meanwhile, the investigators evaluate the effect of tES on electroencephalography (EEG) of both resting and task-related signal. The hypothesis of this study is that tES can improve the cognitive function of emotion by modulating brain activity.

DETAILED DESCRIPTION:
This is a randomized, single-blind, sham-controlled study using transcranial Electrical Stimulation (tES) for 7-day treatment. Participants were randomly assigned to transcranial alternating current stimulation (tACS) group, transcranial direct current stimulation (tDCS) group or sham-control group. Active tES comprised 20 min sessions of 1.5 mA peak-to-peak current delivered over the dorsolateral prefrontal cortex, for 7 consecutive days. Sham group was administered similarly, but with current turned off after 30s. Apart from studying the effects of tES on physiology signals, subjective scale assessments and behavioral data are performed before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* with normal or corrected to normal vision
* participant or guardian need to sign informed consent

Exclusion Criteria:

* reported neurological or psychiatric disorders
* history of any form of transcranial electrical stimulation experience
* use of mood stabilizer
* history of substance abuse or dependence
* severe somatic diseases that might interfere with regular antidepressant treatment including conditions such as kidney and liver failure, uncontrolled hypertension, cardiovascular, cerebrovascular and pulmonary disease, thyroid disease, diabetes, epilepsy and asthma
* use of anti-inflammatory medication for longer than 7 days in the last two months preceding the trial
* use of immunosuppressive medication such as oral steroid hormones women in pregnancy or lactation period

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The change of event-related potentials (ERPs) before and after stimulation. | Day1, Day7
  The aim is to explore whether tES have a regulation effect on emotion processing of dynamic course. In the task, participants need to concentrate on the emotional picture with positive, negative and neutral faces. Then, different ERP components elicited by positive, negative and neutral faces using the signals recorded during facial emotion identification task. The investigators will analyze the ERP components change before and after stimulation to access tES effect on emotion processing.
The change of resting EEG power and lateralization index before and after stimulation. | Day1, Day7
  The aim is to explore whether tES have a regulation effect at-risk of frequency domain. In the resting task, 8 mins resting EEG will be recorded. During recording, participants need to remain still and relaxed with their eyes open (O) and closed (C) in two alternating orders. In order to access tES effect on resting EEG, spectral analysis will be executed after the experiment. Analysis in frequency domain also contributed to expound the brain mechanism related cerebral cortex in emotion processing. In specific, EEG power of delta, theta, alpha, beta and gamma band would be calculated after recording. Besides, the EEG lateralization index also be analyzed between left and right brain.

SECONDARY OUTCOMES:
The change of scores in subjective scale measurement of State-Trait Anxiety Inventory from pre- to post-stimulation. | Day1, Day7
  The main objective is to explore whether tES has an effect on subjective scale after stimulation. The scales include State-Trait Anxiety Inventory (STAI) and Difficulties in Emotion Regulation Scale (DERS). The STAI is a brief self-report assessment for trait anxiety and state measurement. The scales contain two 20-item pools of emotional state and personality trait, each item rated on a 4-point intensity scale ranging from not at all to very much so or from never to almost always respectively. DERS, on the other hand, is also a self-report measure function to assess the emotion regulation.
The change of scores in subjective scale measurement of Difficulties in Emotion Regulation Scale (DERS) from pre- to post-stimulation. | Day1, Day7
  The main objective is to explore whether tES has an effect on subjective scale after stimulation. Difficulties in Emotion Regulation Scale (DERS), which is also a self-report measure function to assess the emotion regulation.
The change of behavioral data from pre- to post-stimulation. | Day1, Day7
  The aim is to explore whether tES have a regulation effect on emotion identification task. During the task, participants need to respond as quickly as probable to emotional stimuli by pressing the space bar. Reaction time and accuracy from the facial emotion identification task pre- and post-stimulation would be recorded. After the experiment, the investigators will access the stimulation effect on their behavioral data change.
Adverse events from baseline to Day1. | Day2, Day3, Day4, Day5, Day6, Day7
  The aim is to evaluate the adverse effects during the stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China